CLINICAL TRIAL: NCT00351598
Title: Tumour Volume as an Independent Prognostic Factor in Patients With Non-Small Cell Lung Cancer - A Protocol for a Prospective Database.
Brief Title: Lung Tumour Volume Database
Status: Completed | Type: Observational
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: TROG 99.05
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tumour Volume; Prognostic value
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with loco-regional, NSCLC treated by definitive radiotherapy.
  Interventions: Radiation: Definitive Radiotherapy

INTERVENTIONS:
Radiation: Definitive Radiotherapy — 60Gy in 6 weeks, 50Gy in 4 weeks. Each individual fraction should not exceed 2.5Gy.
  Other Names: Radiation

SUMMARY:
The main aim is to determine, in patients with locoregional, non-small cell lung cancer (NSCLC) treated by definitive radiotherapy, the influence on survival of the volume of primary tumour, as measured from CT imaging, after adjusting for the effect of the current TNM staging system and other known prognostic factors (especially ECOG performance and weight loss).

DETAILED DESCRIPTION:
Patients with locoregional non small cell lung cancer are registered on study after tumour volumes are outlined by a radiologist and prior to the commencement of any treatment.

All patients must have recorded the volume of disease in the primary tumour (and of involved nodes > 1 cm diameter) as measured from a CT scan performed according to a standard set of conditions.

Following registration patients are treated with Definitive radiotherapy with or without chemotherapy. Follow-up will occur with the collection of a minimum amount of data every 12 months from the date of registration on study.

Quality Assurance procedures will be implemented with each site that participates in the study.

ELIGIBILITY:
Inclusion Criteria:

Must satisfy ALL of the following

* NSCLC - histological or cytological diagnosis of non-small cell lung cancer
* Intra-thoracic disease - disease is confined to the primary site, with or without intrathoracic lymph nodes
* CT planning - CT imaging of the thorax has been performed as part of the planning procedure
* Definitive radiotherapy - it is planned to give definitive radiotherapy with or without chemotherapy (prior to, during or after radiotherapy). Definitive radiotherapy is defined as 60 Gy in 6 weeks, 50 Gy in 4 weeks or at least the equivalent of either of these. The size of each individual; fraction should not exceed 2.5 Gy.
* Measurable disease - the primary tumour and nodes with maximum diameter greater than 1cm represent measurable disease

Exclusion Criteria:

A patient satisfying ANY of the following is ineligible

* Symptomatic or radiological evidence of metastatic disease
* Prior treatment for non-small cell lung cancer
* Surgical resection is part of initial treatment
* Palliative radiotherapy planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with loco-regional non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 531 (Actual)
Dates: Start 1999-09; Primary Completion 2009-02 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Survival | End of Study
  Survival duration defined as the time from date of registration until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: David Ball, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (15):
- Australia (13):
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Mater QRI, South Brisbane, Queensland
  - East Coast Cancer Centre, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Auckland Hospital, Auckland, New Zealand
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Result] Ball DL, Fisher R, Burmeister B, Graham P, Joseph D, Penniment M, Krawitz H, Wheeler G, Poulsen M, Vinod S, McClure B. Stage is not a reliable indicator of tumor volume in non-small cell lung cancer: a preliminary analysis of the Trans-Tasman Radiation Oncology Group 99-05 database. J Thorac Oncol. 2006 Sep;1(7):667-72. PMID 17409934
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au